CLINICAL TRIAL: NCT04377165
Title: Innovative Tool to Limit Spread of COVID 19 in Residential Aged Care
Brief Title: Innovative Tool to Limit Spread of COVID 19 in Residential Aged Care Facilities
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Engagement issues, poor recruitment to study
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Care Collective Study
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-04

CONDITIONS: COVID; Influenza; Gastroenteritis
Keywords: Infection Control
MeSH Terms: conditions — Influenza, Human; Gastroenteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newsfeed (Active Comparator): This will provide you with reliable accurate information on the pandemic.
  Interventions: Behavioral: Newsfeed function
- Gamification (Experimental): The gamification function will allow users to earn points for actions completed. The gamification function has links to resources for infection control, watching or completing tasks or playing games to earn points. Points can be viewed at a facility level, state level or national level.
  Interventions: Behavioral: Gamification

INTERVENTIONS:
Behavioral: Gamification — This will provide the user with the newsfeed function and the addition of a gamification function
  Arms: Gamification
Behavioral: Newsfeed function — This will provide the user with reliable accurate information on the pandemic.
  Arms: Newsfeed

SUMMARY:
This project is a randomised trial in order to determine if "gamification" can result in behaviour change for healthcare workers in the residential aged care setting. The app is for Age Care and care workers at the front line who are working to protect those most vulnerable to COVID-19. There are 2 groups in this trial on group will receive current and accurate information from an app. The other group will receives the app with the addition of a gamification competent, this will include rewarding experiences for staff doing safety behaviours and wellbeing behaviours. The purpose of the gamification is to create a calming and reassuring experience that injects positivity and joy where possible during this stressful time.

DETAILED DESCRIPTION:
The study design will be a multi- centre cluster randomised control trial, where Age Care facilities are randomised into two groups:

1. Newsfeed- gets the app with newsfeed only
2. Gamification group- gets the full gamified app, including the newsfeed Workers in our network of residential aged care facilities will be invited to participate in a study of communication of information regarding COVID-19 and how they will play a role in preventing its spread.

ELIGIBILITY:
Inclusion Criteria:

* Age Health Care Worker

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
To compare the hours of sick leave used over the course of the 4-week period post randomisation for each group | 4 weeks
  Compare the number of sick leave prior to users utilising the app and at the end of the 4 weeks between the arms

SECONDARY OUTCOMES:
To compare handwashing behaviour | 4 weeks
  Compare the amount of soap/sanitiser used between the arms
To compare self-testing rates | 4 weeks
  Compare the number of self tests between the two arms
To compare the level of surface wipe down | 4 weeks
  Compare the amount of wipes/disinfectant used between the two arms
To compare number of COVID-19 tests completed in Facilities | 4 weeks
  Compare the number of COVID-19 tests between the two arms
To compare the number of COVID 19 infections in facilities | 4 weeks
  Compare the number of COVID-19 infections between the arms
To compare the other types of outbreaks (Flu, gastroenteritis) | 4 weeks
  Compare the number of flu and gastroenteritis outbreaks between the arms
To compare the awareness of COVID 19 training available to workers in the facilities | 4 weeks
  Compare the COVID 19 training between the two arms, this is via a self reported survey
To compare the awareness of PPE training available to workers in the facilities | 4 weeks
  Compare the awareness of PPE training of the workers in the two arms, this is captured in self reported survey
To compare the levels of PPE material used in | 4 weeks
  Compare the amount of PPE used between the arms
To compare the wellbeing and self-efficacy of the two groups | 4 weeks
  Compare the wellbeing and self-efficacy between the two arms, this is captured in a self reported survey.

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, PhD, Principal Investigator — The University of Queensland

IPD SHARING:
Plan to Share IPD: No